CLINICAL TRIAL: NCT03093324
Title: A Phase 3 Study in Subjects With Relapsing Remitting Multiple Sclerosis to Evaluate the Tolerability of ALKS 8700 and Dimethyl Fumarate
Brief Title: A Tolerability Study of ALKS 8700 in Subjects With Relapsing Remitting Multiple Sclerosis (RRMS) EVOLVE-MS-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK8700-A302; 2017-001294-16 (EudraCT Number)
Record Dates: First submitted 2017-03-16; First posted 2017-03-28 (Actual); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: RRMS; Multiple Sclerosis; MS; Alkermes; ALKS 8700; Dimethyl Fumarate; DMF; Tecfidera
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALKS 8700 (Experimental): Oral capsules, administered orally twice daily.
  Interventions: Drug: ALKS 8700
- Dimethyl Fumarate (Active Comparator): Oral capsules, administered orally twice daily.
  Interventions: Drug: Dimethyl Fumarate

INTERVENTIONS:
Drug: ALKS 8700 — Administered as specified in the treatment arm.
  Arms: ALKS 8700
Drug: Dimethyl Fumarate — Administered as specified in the treatment arm.
  Other Names: Tecfidera
  Arms: Dimethyl Fumarate

SUMMARY:
The objectives of this study are to evaluate the utility of two gastrointestinal (GI) symptom scales (Individual GI Symptom and Impact Scale {IGISIS} and Global GI Symptom and Impact Scale {GGISIS}) in assessing GI tolerability in adult subjects with RRMS after administration of ALKS 8700 or Dimethyl Fumarate (DMF) in Part A, to compare the GI tolerability of ALKS 8700 and DMF in adult subjects with RRMS using IGISIS and GGISIS in Part B, and to Evaluate the safety and tolerability of ALKS 8700 in adult subjects with RRMS in Parts A and B.

ELIGIBILITY:
Key Inclusion Criteria:

* Capable of understanding and complying with the protocol
* Has a confirmed diagnosis of RRMS
* Neurologically stable with no evidence of relapse within 30 days prior to randomization
* Agrees to use an acceptable method of contraception for the duration of the study and for 30 days after any study drug administration, or is surgically sterile or post-menopausal

Key Exclusion Criteria:

* Have any finding(s) that would compromise the safety of the subject, affect the subject's ability to adhere to the protocol visit schedule or to fulfill visit requirements, or would make the subject unsuitable for participation in the study
* Diagnosis of primary progressive, secondary progressive, or progressive relapsing MS
* History of clinically significant cardiovascular, pulmonary, GI, dermatologic, psychiatric, neurologic (other than MS), endocrine, renal, and/or other major disease that would preclude participation in a clinical trial
* History of GI surgery (except appendectomy that occurred more than 6 months prior to screening
* History of clinically significant recurring or active gastrointestinal symptoms (eg, nausea, diarrhea, dyspepsia, constipation) within 3 months of screening
* Chronic use (7 days) of medical therapy to treat any GI symptoms within 1 month of screening Has a clinically significant medical condition or observed abnormality at screening
* History of a myocardial infarction, including a silent myocardial infarction or unstable angina
* History of clinically significant drug or alcohol abuse within the past year prior to screening
* Clinically significant history of suicidal ideation or suicidal behavior in the last 12 months
* Subject is pregnant or breastfeeding or plans to become pregnant or begin breastfeeding at any point during the study and for 30 days after any study drug administration
* Prior use of Dimethyl Fumarate (DMF)

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (60):
- United States (50):
  - Alkermes Investigational Site, Cullman, Alabama
  - Alkermes Investigational Site, Phoenix, Arizona
  - Alkermes Investigational Site, Tucson, Arizona
  - Alkermes Investigational Site, Long Beach, California
  - Alkermes Investigational Site, San Diego, California
  - Alkermes Investigational Site, Basalt, Colorado
  - Alkermes Investigational Site, Centennial, Colorado
  - Alkermes Investigational Site, Denver, Colorado
  - Alkermes Investigational Site, Middlebury, Connecticut
  - Alkermes Investigational Site, Stamford, Connecticut
  - Alkermes Investigational Site, Washington D.C., District of Columbia
  - Alkermes Investigational Site, Atlantis, Florida
  - Alkermes Investigational Site, Bradenton, Florida
  - Alkermes Investigational Site, Maitland, Florida
  - Alkermes Investigational Site, Naples, Florida
  - Alkermes Investigational Site, Ormond Beach, Florida
  - Alkermes Investigational Site, Sarasota, Florida
  - Alkermes Investigational Site, Tampa, Florida
  - Alkermes Investigational Site, Vero Beach, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Columbus, Georgia
  - Alkermes Investigational Site, Evanston, Illinois
  - Alkermes Investigational Site, Des Moines, Iowa
  - Alkermes Investigational Site, Lenexa, Kansas
  - Alkermes Investigational Site, Alexandria, Louisiana
  - Alkermes Investigational Site, Detroit, Michigan
  - Alkermes Investigational Site, Golden Valley, Minnesota
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Albuquerque, New Mexico
  - Alkermes Investigational Site, Patchogue, New York
  - Alkermes Investigational Site, Stony Brook, New York
  - Alkermes Investigational Site, Syracuse, New York
  - Alkermes Investigational Site, Charlotte, North Carolina
  - Alkermes Investigational Site, Greensboro, North Carolina
  - Alkermes Investigational Site, Winston-Salem, North Carolina
  - Alkermes Investigational Site, Canton, Ohio
  - Alkermes Investigational Site, Columbus, Ohio
  - Alkermes Investigational Site, Dayton, Ohio
  - Alkermes Investigational Site, Oklahoma City, Oklahoma
  - Alkermes Investigational Site, Charleston, South Carolina
  - Alkermes Investigational Site, Greer, South Carolina
  - Alkermes Investigational Site, Old Point Station, South Carolina
  - Alkermes Investigational Site, Spartanburg, South Carolina
  - Alkermes Investigational Site, Franklin, Tennessee
  - Alkermes Investigational Site, Knoxville, Tennessee
  - Alkermes Investigational Site, Dallas, Texas
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, Newport News, Virginia
  - Alkermes Investigational Site, Richmond, Virginia
  - Alkermes Investigational Site, Seattle, Washington
- Germany (4):
  - Alkermes Investigational Site, Dresden
  - Alkermes Investigational Site, Leipzig
  - Alkermes Investigational Site, Ulm
  - Alkermes Investigational Site, Westerstede
- Poland (6):
  - Alkermes Investigational Site, Gdansk
  - Alkermes Investigational Site, Katowice
  - Alkermes Investigational Site, Kielce
  - Alkermes Investigational Site, Lodz
  - Alkermes Investigational Site, Plewiska
  - Alkermes Investigational Site, Szczecin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bowen JD, Stulc J, Hunter SF, Chen H, Lewin JB, Scaramozza M, Bozin I, Then Bergh F. Diroximel Fumarate in Patients with Relapsing-Remitting Multiple Sclerosis: NEDA-3 After Re-Baselining in the Phase 3 EVOLVE-MS-1 Study. Adv Ther. 2024 Aug;41(8):3396-3406. doi: 10.1007/s12325-024-02901-1. Epub 2024 Jun 15. PMID 38878121
- [Derived] Wundes A, Wray S, Gold R, Singer BA, Jasinska E, Ziemssen T, de Seze J, Repovic P, Chen H, Hanna J, Messer J, Miller C, Naismith RT. Improved gastrointestinal profile with diroximel fumarate is associated with a positive impact on quality of life compared with dimethyl fumarate: results from the randomized, double-blind, phase III EVOLVE-MS-2 study. Ther Adv Neurol Disord. 2021 Mar 19;14:1756286421993999. doi: 10.1177/1756286421993999. eCollection 2021. PMID 33796143
- [Derived] Naismith RT, Wundes A, Ziemssen T, Jasinska E, Freedman MS, Lembo AJ, Selmaj K, Bidollari I, Chen H, Hanna J, Leigh-Pemberton R, Lopez-Bresnahan M, Lyons J, Miller C, Rezendes D, Wolinsky JS; EVOLVE-MS-2 Study Group. Diroximel Fumarate Demonstrates an Improved Gastrointestinal Tolerability Profile Compared with Dimethyl Fumarate in Patients with Relapsing-Remitting Multiple Sclerosis: Results from the Randomized, Double-Blind, Phase III EVOLVE-MS-2 Study. CNS Drugs. 2020 Feb;34(2):185-196. doi: 10.1007/s40263-020-00700-0. PMID 31953790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 70 investigative sites in the United States (US), Germany, and Poland from March 15, 2017 to June 27, 2019.
Pre-assignment Details: A total of 506 participants with relapsing remitting multiple-sclerosis were enrolled in this study. Of which 504 participants received study drug and randomized in Parts A and B of the study (253 participants in ALKS 8700 group and 251 in Dimethyl Fumarate group). A total of 478 participants completed the study.
Groups:
- ALKS 8700: Participants received ALKS 8700 231 milligrams (mg) along with ALKS 8700-matching placebo, oral capsules, twice daily (BID), for Week 1, followed by administration of ALKS 8700 462 mg, oral capsules, BID, for Week 2 to 5.
- Dimethyl Fumarate (DMF): Participants received DMF 120 mg along with DMF-matching placebo, oral capsules, BID for Week 1, followed by administration of DMF 240 mg and DMF-matching placebo, oral capsules, BID, for week 2 to 5.
Period: Overall Study
Arm/Group | ALKS 8700 | Dimethyl Fumarate (DMF)
Started (All enrolled participants.) | 254 | 252
Safety Population (All enrolled participants who received at least one dose of study drug.) | 253 | 251
Completed | 245 | 233
Not Completed | 9 | 19
Not completed — Adverse Event | 4 | 15
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Deviation | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: The Safety population included all enrolled participants who had received at least one dose of study drug during the double-blind Treatment Period.
Groups:
- Total: Total of all reporting groups
Arm/Group | ALKS 8700 | Dimethyl Fumarate (DMF) | Total
Number analyzed (Participants) | 253 | 251 | 504
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (10.96) | 43.7 (9.90) | 43.7 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 190 | 367
  Male | 76 | 61 | 137
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 248 | 241 | 489
  Hispanic or Latino | 5 | 10 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 232 | 227 | 459
  Black or African American | 20 | 20 | 40
  Other | 0 | 2 | 2
  Asian | 0 | 1 | 1
  Multiple races | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Days With Any Individual Gastrointestinal Symptom and Impact Scale (IGISIS) Individual Symptom Intensity Score ≥2 Relative to Exposure Days in Parts A and B
Description: IGISIS assessed the intensity of five individual GI symptoms: nausea, vomiting, upper abdominal pain, lower abdominal pain, and diarrhea. Participants rated the intensity of each individual symptom via an 11-point numeric rating scale ranging from 0 (did not have) to 10 (extreme). IGISIS was completed by the participants using e-diaries.
Time Frame: End of treatment (up to Week 6) for both Parts A and B
Population: The full analysis set (FAS) population included all enrolled participants in the Safety population who had at least one postbaseline GI tolerability assessment (such as IGISIS) on or before the last dose date.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ALKS 8700 | Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 253 | 249
days | 1.5 (2.85) | 2.5 (4.68)
Statistical Analysis 1: Comparison: ALKS 8700 vs Dimethyl Fumarate (DMF); Number of event days was analyzed by a negative binomial regression model, with the logarithmic transformation of the number of exposure days as the ''offset'' parameter and treatment group as a factor and adjusting for study part, region (US and non-US), age, and body mass index (BMI); Test type: Superiority; p = 0.0003, Negative Binomial Regression Model; Rate ratio = 0.542, 95% CI 2-sided [0.390 to 0.754]

2. Secondary Outcome: Number of Days With Any IGISIS Individual Symptom Intensity Score ≥2 Relative to Exposure Days in Part B
Description: as for outcome 1
Time Frame: End of treatment (up to Week 6) for Part B
Population: The FAS population included all enrolled participants in the Safety population who had at least one postbaseline GI tolerability assessment (such as IGISIS) on or before the last dose date. Number analyzed are the participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ALKS 8700 | Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 253 | 249
days | 1.3 (2.70) | 2.2 (4.22)
Statistical Analysis 1: Comparison: ALKS 8700 vs Dimethyl Fumarate (DMF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0007, Negative Binomial Regression Model; Rate ratio = 0.520, 95% CI 2-sided [0.356 to 0.760]

3. Secondary Outcome: Number of Days With Any IGISIS Individual Symptom Intensity Score ≥1 Relative to Exposure Days in Parts A and B
Description: as for outcome 1
Time Frame: End of treatment (up to Week 6) for both Parts A and B
Population: The FAS population included all enrolled participants in the Safety population who had at least one postbaseline GI tolerability assessment (such as IGISIS) on or before the last dose date.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ALKS 8700 | Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 253 | 249
days | 2.9 (4.46) | 3.9 (5.84)
Statistical Analysis 1: Comparison: ALKS 8700 vs Dimethyl Fumarate (DMF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.009, Negative Binomial Regression Model; Rate ratio = 0.714, 95% CI 2-sided [0.554 to 0.921]

4. Secondary Outcome: Number of Days With Any IGISIS Individual Symptom Intensity Score ≥3 Relative to Exposure Days in Parts A and B
Description: as for outcome 1
Time Frame: End of treatment (up to Week 6) for both Parts A and B
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ALKS 8700 | Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 253 | 249
days | 0.9 (2.25) | 1.5 (3.85)
Statistical Analysis 1: Comparison: ALKS 8700 vs Dimethyl Fumarate (DMF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.009, Negative Binomial Regression Model; Rate ratio = 0.555, 95% CI 2-sided [0.357 to 0.862]

5. Secondary Outcome: Number of Days With a Global GI Symptom and Impact Scale (GGISIS) Symptom Intensity Score ≥1 Relative to Exposure Days in Parts A and B
Description: GGISIS is a global scale to assess the overall intensity of GI symptoms (nausea, vomiting, upper abdominal pain, lower abdominal pain, and diarrhea). Participants rated the intensity of GI symptoms via an 11-point numeric rating scale ranging from 0 (did not have) to 10 (extreme). GGISIS was completed by the participants using e-diaries.
Time Frame: End of treatment (up to Week 6) for both Parts A and B
Population: The FAS population included all enrolled participants in the Safety population who had at least one postbaseline GI tolerability assessment (such as GGISIS) on or before the last dose date. Number analyzed are the participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ALKS 8700 | Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 253 | 249
days | 2.1 (4.43) | 2.8 (5.19)
Statistical Analysis 1: Comparison: ALKS 8700 vs Dimethyl Fumarate (DMF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.033, Negative Binomial Regression Model; Rate ratio = 0.696, 95% CI 2-sided [0.499 to 0.972]

6. Secondary Outcome: Number of Days With a GGISIS Symptom Intensity Score ≥2 Relative to Exposure Days in Parts A and B
Description: as for outcome 5
Time Frame: End of treatment (up to Week 6) for both Parts A and B
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ALKS 8700 | Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 253 | 249
days | 1.1 (3.25) | 1.5 (3.53)
Statistical Analysis 1: Comparison: ALKS 8700 vs Dimethyl Fumarate (DMF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.068, Negative Binomial Regression Model; Rate ratio = 0.662, 95% CI 2-sided [0.425 to 1.031]

7. Secondary Outcome: Number of Days With a GGISIS Symptom Intensity Score ≥3 Relative to Exposure Days in Parts A and B
Description: as for outcome 5
Time Frame: End of treatment (up to Week 6) for both Parts A and B
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ALKS 8700 | Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 253 | 249
days | 0.7 (2.26) | 0.9 (2.57)
Statistical Analysis 1: Comparison: ALKS 8700 vs Dimethyl Fumarate (DMF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.215, Negative Binomial Regression Model; Rate ratio = 0.713, 95% CI 2-sided [0.417 to 1.217]

8. Secondary Outcome: Worst IGISIS Individual Symptom Intensity Score During the 5-Week Treatment Period in Parts A and B
Description: IGISIS assessed the intensity of five individual GI symptoms: nausea, vomiting, upper abdominal pain, lower abdominal pain, and diarrhea. Participants rated the intensity of each individual symptom via an 11-point numeric rating scale ranging from 0 (did not have) to 10 (extreme). IGISIS was completed by the participants using e-diaries. Scores were averaged for 5-week treatment period.
Time Frame: End of treatment (up to Week 6) for both Parts A and B
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ALKS 8700 | Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 253 | 249
score on a scale
  Nausea | 0.9 (1.55) | 1.2 (1.98)
  Vomiting | 0.2 (0.74) | 0.6 (1.84)
  Upper Abdominal Pain | 0.8 (1.58) | 1.3 (2.06)
  Lower Abdominal Pain | 0.8 (1.60) | 1.0 (1.84)
  Diarrhea | 1.1 (2.09) | 1.3 (2.19)
Statistical Analysis 1: Comparison: ALKS 8700 vs Dimethyl Fumarate (DMF); Nausea: DMF is used as a referenced group in the model, adjusting for study parts, region (US and non-US), age and BMI; Test type: Superiority; p = 0.043, ANCOVA; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-0.6 to -0.0], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: ALKS 8700 vs Dimethyl Fumarate (DMF); Vomiting: DMF is used as a referenced group in the model, adjusting for study parts, region (US and non-US), age and BMI; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: ALKS 8700 vs Dimethyl Fumarate (DMF); Upper Abdominal Pain: DMF is used as a referenced group in the model, adjusting for study parts, region (US and non-US), age and BMI; Test type: Superiority; p = 0.001, ANCOVA; Least Squares Mean Difference = -0.5, 95% CI 2-sided [-0.9 to -0.2], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: ALKS 8700 vs Dimethyl Fumarate (DMF); Lower Abdominal Pain: DMF is used as a referenced group in the model, adjusting for study parts, region (US and non-US), age and BMI; Test type: Superiority; p = 0.403, ANCOVA; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-0.4 to 0.2], Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: ALKS 8700 vs Dimethyl Fumarate (DMF); Diarrhea: DMF is used as a referenced group in the model, adjusting for study parts, region (US and non-US), age and BMI; Test type: Superiority; p = 0.261, ANCOVA; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.2], Standard Error of Mean 0.19

9. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: End of study (up to Week 10)
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | ALKS 8700 | Dimethyl Fumarate (DMF)
Number analyzed (Participants) | 253 | 251
participants | 198 | 210

ADVERSE EVENTS:
Time Frame: End of study (up to Week 10)
Description: The Safety population included all enrolled participants who had received at least one dose of study drug during the double-blind Treatment Period.
Arm/Group | ALKS 8700 | Dimethyl Fumarate (DMF)
All-Cause Mortality (participants affected / at risk) | 0/253 | 0/251
Serious Adverse Events (participants affected / at risk) | 4/253 | 3/251
Other Adverse Events (participants affected / at risk) | 175/253 | 191/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALKS 8700 (N=253) | Dimethyl Fumarate (DMF) (N=251)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 3 | 2
Suicide attempt (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALKS 8700 (N=253) | Dimethyl Fumarate (DMF) (N=251)
Abdominal pain (Gastrointestinal disorders) | 16 | 24
Abdominal pain lower (Gastrointestinal disorders) | 15 | 17
Abdominal pain upper (Gastrointestinal disorders) | 17 | 39
Diarrhoea (Gastrointestinal disorders) | 39 | 56
Nausea (Gastrointestinal disorders) | 37 | 52
Vomiting (Gastrointestinal disorders) | 9 | 22
Fatigue (General disorders) | 6 | 13
Feeling hot (General disorders) | 4 | 6
Nasopharyngitis (Infections and infestations) | 15 | 11
Upper respiratory tract infection (Infections and infestations) | 9 | 9
Urinary tract infection (Infections and infestations) | 8 | 9
Alanine aminotransferase increased (Investigations) | 14 | 9
Aspartate aminotransferase increased (Investigations) | 9 | 5
Urine albumin/creatinine ratio increased (Investigations) | 6 | 2
Headache (Nervous system disorders) | 10 | 14
Multiple sclerosis relapse (Nervous system disorders) | 8 | 5
Erythema (Skin and subcutaneous tissue disorders) | 20 | 21
Generalised erythema (Skin and subcutaneous tissue disorders) | 4 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 18
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 6
Rash (Skin and subcutaneous tissue disorders) | 4 | 6
Flushing (Vascular disorders) | 83 | 102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT03093324/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT03093324/SAP_001.pdf